CLINICAL TRIAL: NCT06227169
Title: From Court to the Community: Improving Access to Evidence-Based Treatment for Underserved Justice-Involved Youth At-Risk for Suicide
Brief Title: From Court to the Community
Acronym: JJ-COPES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kathleen Kemp, Research Psychologist, Rhode Island Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 201922; R01MH129770 (NIH)
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Thoughts and Behaviors
MeSH Terms: conditions — Suicidal Ideation; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community mental health clinician training cohort 1 (Experimental): In this stepped wedge design, cohorts of community-based clinicians receive a training in how to conduct an evidence-based cognitive behavioral intervention in suicide prevention for justice-involved youth. There are 15 clinicians in each training cohort.
  Interventions: Behavioral: JJ-COPES Training
- Community mental health clinician training cohort 2 (Experimental): In this stepped wedge design, cohorts of community-based clinicians receive a training in how to conduct an evidence-based cognitive behavioral intervention in suicide prevention for justice-involved youth. There are 15 clinicians in each training cohort.
  Interventions: Behavioral: JJ-COPES Training
- Community mental health clinician training cohort 3 (Experimental): In this stepped wedge design, cohorts of community-based clinicians receive a training in how to conduct an evidence-based cognitive behavioral intervention in suicide prevention for justice-involved youth. There are 15 clinicians in each training cohort.
  Interventions: Behavioral: JJ-COPES Training

INTERVENTIONS:
Behavioral: JJ-COPES Training — • The JJ-COPES training is derived from an empirically supported CBT manual designed for outpatient treatment of suicidal adolescents. JJ-COPES training focuses on teaching 4 primary treatment strategies plus a caregiver session to community-based clinicians.

SUMMARY:
Youth involved in the juvenile justice system evidence disproportionately high rates of suicidal thoughts and behavior (STB) and non-suicidal self-injury (NSSI) compared to adolescents in the general population. It is estimated that upwards of 50% of justice-involved youth (JIY) in secure facilities report NSSI and suicide attempts.1-3 Suicide attempts are estimated to be between two and four times more frequent in incarcerated JIY than adolescents in the community,4 and the rates of STB in JIY are higher than non-JIY in the community. The overwhelming majority of JIY are not placed in secure facilities and almost all incarcerated youth are eventually released to the community.5 Consequently, STB is a major concern of JIY residing in the community and it is critical that this population has access to evidence-based treatment for STB and NSSI. Contributing to the problem, racial and ethnic minority youth are disproportionately represented among JIY6 and JIY are more likely to reside in neighborhoods with limited resources,7 including restricted access to community mental health treatment.8,9 Further, most community mental health providers who treat JIY have not been trained in evidence-based interventions that are specifically designed to treat NSSI and STB; this often leads to JIY experiencing prolonged periods of NSSI and/or STB.10 Training community mental health providers who serve JIY in the detection and treatment of NSSI and STB has promise to decrease the overall suicide risk for JIY. The primary goal of this application is to train community providers in established, core strategies for adolescent STB and NSSI.11 The training program has been used in two clinical trials, refined for inpatient psychiatric and Emergency Department providers, and modified for use in community practice.

Our Primary Aim is to implement a systems-level intervention focused on increasing access to evidence-based treatment strategies specifically designed to treat STB and NSSI behaviors for the JIY referred to outpatient care by the RIFC. First, the investigators will conduct a stepped wedge cluster randomized trial with 9 Rhode Island CMHAs who serve JIY. After all sites complete a Usual Care phase, three CMHAs per year will be randomized to the Preparation Phase to receive training in evidence-based strategies for NSSI and STB, using a training program called COPES,11 developed by the MPI for inpatient psychiatry units and Emergency Departments, transported to CMHAs by Consultant and consistent with recommendations in SAMHSA's Youth Suicide Treatment Guide.13 Agencies then move into Implementation Phase for consultation and support followed by a Sustainment phase. Second, guided by the Reach Effectiveness-Adoption Implementation Maintenance (RE-AIM) framework, the investigators will conduct qualitative interviews and administer agency and provider demographic questionnaires and organizational readiness measures with CMHA providers and administrators to identify system-, agency-, and provider-level factors that promote or hinder the uptake and sustainment of evidence-based treatment for STB and NSSI at CMHAs serving JIY. At the provider level, the investigators hypothesize that training in the use of evidence-based treatment strategies for STB and NSSI will: a) significantly increase the use of these strategies and b) the quality of their delivery will be in the "acceptable" range during the Sustainment Phase. At the client/patient level, the investigators hypothesize that the intervention will keep families engaged more than Usual Care phase, increase sessions attended, and reduce rates of adolescent STB and NSSI that require emergency psychiatric care. At the systems level, the investigators hypothesize that the training program will be sustained for at least one year, and up to 3 years, by CMHA administrators. The investigators will also examine factors that may affect the effectiveness of uptake and sustainment of the training program, i.e., organizational readiness, climate, and leadership at each CMHA.

ELIGIBILITY:
Inclusion Criteria:

* Eligible providers must have active caseloads of justice-involved youth, be willing to be trained in COPES, and participate in implementation efforts

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Electronic Medical Record | 54 months
  Therapy notes will be coded for evidence of provider-level outcomes, including: (1) use of general techniques consistent with cognitive-behavioral therapy and (2) use of specific JJ COPES + skills (e.g., safety plan), as well as patient-level outcomes, including: (3) treatment attendance; (4) emergency/crisis service use for STB/NSSI; (5) instances of self-injury; and (6) evidence of suicidal thoughts or attempts

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No